CLINICAL TRIAL: NCT00442910
Title: Phase 1 Study of the Safety and Acceptability of 3% w/w SPL7013 Gel (VivaGel™) Applied Vaginally in Sexually Active Young Women
Brief Title: Safety and Acceptability of SPL7013 Gel (VivaGel™) in Sexually Active Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Starpharma Pty Ltd (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Microbicide Trials Network (Network)
Responsible Party: Professor Ian McGowan, Principal Investigator, Microbicide Trials Network
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MTN-004; SPL7013-006
Record Dates: First submitted 2007-03-02; First posted 2007-03-05 (Estimated); Last update posted 2010-06-24 (Estimated); Status verified 2010-06

CONDITIONS: Healthy
Keywords: Safety and Acceptability
MeSH Terms: interventions — astodrimer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 3% SPL7013 (Active Comparator): Intravaginal application of 3.5 g SPL7013 gel twice daily for 14 days
  Interventions: Drug: 3% SPL7013 Gel (VivaGel)
- Placebo for SPL7013 Gel (Placebo Comparator): Intravaginal application of 3.5 g placebo gel twice daily for 14 days
  Interventions: Drug: Placebo Gel
- HEC Placebo Gel (Placebo Comparator): Intravaginal application of 3.5 g HEC placebo gel twice daily for 14 days
  Interventions: Drug: HEC Placebo Gel

INTERVENTIONS:
Drug: 3% SPL7013 Gel (VivaGel) — 3% vaginal gel
  Other Names: VivaGel
  Arms: 3% SPL7013
Drug: Placebo Gel — Placebo for SPL7013 gel
  Arms: Placebo for SPL7013 Gel
Drug: HEC Placebo Gel — HEC Placebo gel intravaginally bd for 14 days
  Other Names: Universal Placebo
  Arms: HEC Placebo Gel

SUMMARY:
There is an urgent need for HIV prevention methods that women can initiate and control themselves. Topical microbicides, substances that kill microbes, represent one such method. The purpose of this study is to assess the safety and to evaluate the acceptability of 3% w/w SPL7013 gel, a topical microbicide, when administered intravaginally for 14 consecutive days in healthy, sexually active HIV uninfected women.

DETAILED DESCRIPTION:
Women continue to comprise a growing proportion of the new HIV infections around the world. A growing body of data suggests that a safe and effective topical microbicide will be a real option of prevention for women in the future. The purpose of this study is to assess the safety and acceptability of 3% SPL7013 Gel when administered intravaginally, twice daily for 14 consecutive days in healthy, sexually-active, HIV-uninfected women.

The expected duration of this study for each participant is 21 days. Study participants will be randomly assigned to one of two arms. Participants in Arm 1 will apply 3.5 g of SPL7013 gel intravaginally twice daily for 14 consecutive days. Participants in Arm 2 will apply a placebo gel intravaginally twice daily for 14 consecutive days. Starpharma produces SPL7013 gel (VivaGel) and will provide it for this study.

After enrollment, participants will attend three study visits. These visits will occur on Days 7, 14, and 21. A follow-up safety visit will occur if necessary. Medical and menstrual history, targeted physical exam, urine and blood collection, cervical swabs, and vaginal smears will occur at all visits. A colposcopy will occur at least once. On Day 2, participants will take part in a phone assessment.

ELIGIBILITY:
Inclusion Criteria:

* HIV-uninfected
* General good health
* Normal Pap result within 12 months prior to study entry
* Predictable menstrual cycle with at least 21 days between menses
* Sexually active
* Willing to use effective methods of contraception for the duration of the study. More information on this criterion can be found in the protocol.
* Willing to abstain from oral-vaginal and penile-anal intercourse for the duration of the study
* Willing to not use other intravaginal products and/or devices for 72 hours prior to study entry through Week 3
* Agree to have partner use condoms provided by study for each act of intercourse during study participation
* Willing to undergo colposcopy if determined necessary by investigator
* Agree to not participate in other drug or device studies during study participation

Exclusion Criteria:

* History of adverse reaction to latex or to any component of the study products
* History of male sex partner having an allergic reaction to latex
* Any abnormal finding on physical or pelvic examination
* Sexually transmitted infection (STI) or reproductive tract infection. More information on this criterion is available in the protocol.
* Diagnosed with STI within 6 months prior to study entry
* Use of oral and/or vaginal preparations of antibiotic or antifungal medications within 30 days prior to study entry
* Gynecological surgical procedure within 90 days prior to study entry
* Certain abnormal laboratory values. More information on this criterion is available in the protocol.
* Received non-therapeutic intravenous drugs within 12 months prior to study entry
* Any social or medical condition, that, in the opinion of the investigator, would interfere with the study
* Pregnant of breastfeeding

Ages: 18 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2007-07; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Incidence of abnormal genital symptoms and/or pelvic exam findings | Throughout study
Occurrence of adverse events and/or abnormal laboratory values | Throughout study

SECONDARY OUTCOMES:
Changes in vaginal microflora | Throughout study
Proportion of participants who report an 80% or greater adherence rate | At Day 7 and Day 14
Proportion of participants who say they would be very likely to use the study product in the future | At Day 14
Reported positive and negative aspects of using study product | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Ian McGowan, MD, PhD, Study Chair — University of California Geffen School of Medicine
Locations (3):
- United States (2):
  - University of South Florida, Tampa, Florida
  - Center for Family Planning Research, Magee-Womens Hospital, Pittsburgh, Pennsylvania
- University of Puerto Rico, San Juan, Puerto Rico

REFERENCES:
- [Background] Balzarini J, Van Damme L. Microbicide drug candidates to prevent HIV infection. Lancet. 2007 Mar 3;369(9563):787-797. doi: 10.1016/S0140-6736(07)60202-5. PMID 17336656
- [Background] Rupp R, Rosenthal SL, Stanberry LR. VivaGel (SPL7013 Gel): a candidate dendrimer--microbicide for the prevention of HIV and HSV infection. Int J Nanomedicine. 2007;2(4):561-6. PMID 18203424
- [Derived] McGowan I, Gomez K, Bruder K, Febo I, Chen BA, Richardson BA, Husnik M, Livant E, Price C, Jacobson C; MTN-004 Protocol Team. Phase 1 randomized trial of the vaginal safety and acceptability of SPL7013 gel (VivaGel) in sexually active young women (MTN-004). AIDS. 2011 May 15;25(8):1057-64. doi: 10.1097/QAD.0b013e328346bd3e. PMID 21505316